CLINICAL TRIAL: NCT00962676
Title: Diagnostic Usefulness of Interferon Gamma Release Assay for Active Tuberculosis in Immunocompromised Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2009-0129
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Tuberculosis
Keywords: suspicious of tuberculosis; immunocompromised patients
MeSH Terms: conditions — Tuberculosis

GROUPS / COHORTS (2):
- immunocompromised group
- non-immunocompromised group

SUMMARY:
For diagnosis of active tuberculosis, interferon-γ release assay based mycobacterium tuberculosis specific antigen may show higher sensitivity than tuberculin skin test in immunocompromised patients. Therefore, interferon-γ release assay have a role as a rapid diagnostic adjunctive methods for active tuberculosis in immunocompromised patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient suspicious of active tuberculosis with immunocompromised condition
* Immunocompromised condition patients with

  1. solid cancer with chemotherapy
  2. hematologic malignancy
  3. organ transplantation
  4. immunosuppressant
  5. ESRD on renal replacement therapy
  6. diabetes
  7. advanced liver cirrhosis

Exclusion Criteria:

* Patients with

  1. less than 20 years
  2. who don't agree the participation of study
  3. hypersensitivity history to tuberculin
  4. pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: suspicious of tuberculosis, immunocompromised patients such cancer patients on chemotherapy, transplantation patients, patients with immunosuppressant
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Univ., Seoul, South Korea